CLINICAL TRIAL: NCT02394015
Title: Multicenter and Retrospective Observational Study to Analyze the Efficacy and Safety of the Combination With Trabectedin and Pegylated Liposomal Doxorubicin (PLD ) in the Treatment of Patients With Platinum-sensitive Recurrent Ovarian Cancer (ROC), According to Data Sheet
Brief Title: Retrospective Study to Analyze the Efficacy and Safety of Trabectedin and Pegylated Liposomal Doxorubicin (PLD ) in the Treatment of Patients With Platinum-sensitive Recurrent Ovarian Cancer (ROC), According to SmPC
Acronym: RETRO-ROC
Status: Completed | Type: Observational
Sponsor: Grupo Español de Investigación en Cáncer de Ovario (Other)
Collaborators: PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: GEICO 1402R; GEI-TRAB-2014-01 (Other: AEMPS)
Record Dates: First submitted 2015-03-10; First posted 2015-03-20 (Estimated); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Epithelial Cancer Recurrent
Keywords: Platinum-sensitive Recurrent Ovarian Cancer
MeSH Terms: interventions — Trabectedin; liposomal doxorubicin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trabectedin+ PLD: Trabectedin and Pegylated Liposomal Doxorubicin (PLD ) in the Treatment of Patients With Platinum-sensitive Recurrent Ovarian Cancer (ROC), according to SmPC.
  Interventions: Drug: Trabectedin and Pegylated Liposomal Doxorubicin

INTERVENTIONS:
Drug: Trabectedin and Pegylated Liposomal Doxorubicin — Trabectedin and Pegylated Liposomal Doxorubicin (PLD ) in the Treatment of Patients With Platinum-sensitive Recurrent Ovarian Cancer (ROC), according to SmPC from October 28, 2009 to October 31, 2014

SUMMARY:
Retrospective Study to Analyze the Efficacy and Safety of Trabectedin and Pegylated Liposomal Doxorubicin (PLD ) in the Treatment of Patients With Platinum-sensitive Recurrent Ovarian Cancer (ROC), According to SmPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received at least one dose of trabectedin - doxorubicin pegylated for recurrent ovarian cancer according to SMPC, between October 28, 2009 and October 31, 2014 and which have not been included in clinical trials where the IMP was trabectedin.

Exclusion Criteria:

* Patients with records unavailable (lost, empty or not recoverable).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have received treatment with trabectedin - DLP for recurrent ovarian cancer according to SMPC, between October 28, 2009 and October 31, 2014 and which have not been included in clinical trials where the IMP was trabectedin.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Efficacy progression-free survival (PFS) | Up to 12 months
  Describe the impact of trabectedin - pegylated liposomal doxorubicin combination of retreatment with platinum ROC, in terms of progression-free survival ( PFS).
Overall survival (OS) | Up to 12 months
  Describe the impact of trabectedin - pegylated liposomal doxorubicin combination of retreatment with platinum ROC, in terms of overall survival (OS ) .

SECONDARY OUTCOMES:
Response rate to previous and post-treatment (Percentage of responses (CR+PR) | Up to 12 months
  Percentage of responses (CR+PR) at pretreatment and post-treatment
Response rate to trabectedin - DLP combination (Percentage of responses (CR+PR) | Up to 12 months
  Percentage of responses ( CR + PR ) to trabectedin - DLP
Clinical Benefit in 4 months (Percentage of clinical benefit (CR + PR + SD) | Up to 12 months
  Percentage of clinical benefit (CR + PR + SD for at least 4 months)
Impact of trabectedin - PLD combination in subsequent treatments | Up to 12 months
  Assessment of the impact of treatment with trabectedin - PLD combination at the beginning of subsequent treatments
Toxicity (adverse events) | Up to 12 months
  type , incidence , severity, frequency, severity and relationship to the treatment of adverse events reported in patients reports
Comparison between PFS and PFS2 | Up to 12 months
  Comparison of the PFS of prior platinum combination TRB + DLP and subsequent platinum PFS.
Hypersensitivity and allergic reactions (Number and Management of hypersensitivity reactions or allergies) | Up to 12 months
  Number and Management of hypersensitivity reactions or allergies.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vidal, MD, Principal Investigator — H. Clinic, Barcelona; Jose M Del Campo, MD, Principal Investigator — H. Vall d'Hebron, Barcelona